CLINICAL TRIAL: NCT05779761
Title: A Randomized Controlled Trial of Brief Interventions for Coping with Distress
Brief Title: Brief Interventions for Coping with Distress
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Teachers College, Columbia University (Other)
Responsible Party: Principal Investigator, Douglas Mennin, Professor of Clinical Psychology, Teachers College, Columbia University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 22-326
Record Dates: First submitted 2023-03-09; First posted 2023-03-22 (Actual); Last update posted 2024-11-21 (Actual); Status verified 2024-11

CONDITIONS: Distress, Emotional; Emotional Dysfunction; Anxiety; Depression
Keywords: Emotion Regulation; Distress Disorders; Anxiety; Depression; Worry; Rumination; Self-Criticism; Skills Training
MeSH Terms: conditions — Anxiety Disorders; Depression; Emotional Regulation; Rumination Syndrome

STUDY DESIGN:
Intervention Model Description: All participants will be randomly assigned to one of three skills trainings for coping with distress.
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Attention Skills Training (Experimental): Participants assigned to Attention Skills Training will receive 6-weeks of self-directed, online skills training on attention regulation skills for coping with distress. Six weekly modules will include 10-15 minutes of narrated videos, as well as suggestions for activities and skills practices between modules. Participants will also schedule weekly, 5-10 minute calls with an assigned skills training coach to discuss the participant's experience with the skills training.
  Interventions: Behavioral: Online, Self-Directed Attention Skills Training with Coaching Support
- Attention and Reflective Thought Skills Training (Experimental): Participants assigned to Attention and Reflective Thought Skills Training will receive 6-weeks of self-directed, online skills training on attention and metacognitive regulation skills for coping with distress. Six weekly modules will include 10-15 minutes of narrated videos, as well as suggestions for activities and skills practices between modules. Participants will also schedule weekly, 5-10 minute calls with an assigned skills training coach to discuss the participant's experience with the skills training.
  Interventions: Behavioral: Online, Self-Directed Attention & Reflective Thought Skills Training with Coaching Support
- Health and Wellness Education Training (Experimental): Participants assigned to Health and Wellness Education Training will receive 6-weeks of self-directed, online skills training on stress-reduction psychoeducation. Six weekly modules will include 10-15 minutes of narrated videos, as well as suggestions for activities and skills practices between modules. Participants will also schedule weekly, 5-10 minute calls with an assigned skills training coach to discuss the participant's experience with the skills training.
  Interventions: Behavioral: Online, Self-Directed Health & Wellness Education Training with Coaching Support

INTERVENTIONS:
Behavioral: Online, Self-Directed Attention Skills Training with Coaching Support — The initial set of modules focus on psychoeducation about distress, the impact that cognitions/behaviors/emotions have on recent situations, and self-monitoring of worry/rumination/self-criticism. The next set of modules focus on the development of attention skills that help regulate one's emotional experience (i.e., recognizing emotions when they are happening, identifying the meaning of a given emotion experience, soothing oneself in the context of negative emotional experiences). All modules will be online and self-directed. An internet-based online platform will be used to promote engagement with and increase accessibility to between-session skills practice and treatment-related activities (e.g., self-monitoring, worksheets). Brief, weekly coaching support (from a trained, masters-level student) will be provided to promote engagement and to help clarify concepts.
  Arms: Attention Skills Training
Behavioral: Online, Self-Directed Attention & Reflective Thought Skills Training with Coaching Support — The initial set of modules focus on psychoeducation about distress, the impact that cognitions/behaviors/emotions have on recent situations, and self-monitoring of worry/rumination/self-criticism. The next set of modules focus on the development of attention and reflective thinking skills that help regulate one's emotional experience (i.e., recognizing emotions when they are happening, identifying the meaning of a given emotion experience, soothing oneself in the context of negative emotional experiences). All modules will be online and self-directed. An internet-based online platform will be used to promote engagement with and increase accessibility to between-session skills practice and treatment-related activities (e.g., self-monitoring, worksheets). Brief, weekly coaching support (from a trained, masters-level student) will be provided to promote engagement and to help clarify concepts.
  Arms: Attention and Reflective Thought Skills Training
Behavioral: Online, Self-Directed Health & Wellness Education Training with Coaching Support — The initial set of modules focus on psychoeducation about stress, the impact that stress has on one's life, and self-monitoring of stress. The next set of modules focus on sleep, time management, nutrition, and exercise. All modules will be online and self-directed. An internet-based online platform will be used to promote engagement with and increase accessibility to between-session skills practice and treatment-related activities (e.g., self-monitoring, worksheets). Brief, weekly coaching support (from a trained, masters-level student) will be provided to promote engagement and to help clarify concepts.
  Arms: Health and Wellness Education Training

SUMMARY:
This study is being done to compare the effectiveness of three different skills trainings to cope with distress. These three trainings are: 1) an attention skills training, 2) an attention and reflective thought skills training, and 3) a health and wellness education training.

DETAILED DESCRIPTION:
Adults living in New York City between the ages of 18-65 and experiencing elevated levels of worry, rumination, and/or self-criticism may be eligible to participate. After being informed about the study and potential risks, participants giving written informed consent will complete an online screening visit to determine full study eligibility. Eligible participant will then be randomized to complete 6-weeks of one of three self-directed, online skills training about coping with distress.

The present study is evaluating whether these skills trainings demonstrate efficacy in: 1) improving outcomes specific to an emotion regulation model of emotional distress (e.g., attentional control, decentering, reappraisal); 2) reducing symptoms of psychological distress (e.g., anxiety, depression, worry, rumination). Primary assessment points will take place before and after the skills training, and will include self-report measures, brief surveys during daily life, as well as computer tasks and measures of brain and body activity (e.g., EEG).

ELIGIBILITY:
Inclusion Criteria:

* Between the ages of 18 and 65
* Fluent in English (and therefore able to provide consent)
* Currently living in New York City
* Access to a smartphone and the internet
* High self-reported worry, rumination, and/or self-criticism
* Meet Diagnostic and Statistical Manual of Mental Disorders - Fifth Edition (DSM-5) criteria for at least one, current psychological disorder

Exclusion Criteria:

* Active suicidal ideation or intent
* Substance dependence disorder, schizophrenia, bipolar-I disorder, or a primary DSM-5 diagnosis of borderline or narcissistic personality disorder
* Individuals currently receiving therapy or psychosocial treatment who do not plan to continue with the same treatment throughout the study period
* Individuals taking psychotropic mediation that has not been stabilized for a period of at least 3 months
* Current students at Teachers College, Columbia University
* Individuals with cardiac conditions, diagnosed hyperhidrosis, and traumatic brain injuries or other neurological conditions (e.g., dementia, Parkinson's, epilepsy)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2023-05-12 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Changes in Ability to Regulate Emotions: Emotion Regulation Questionnaire (ERQ) | Pre-Training, Post-Training (6 weeks after starting the training), and 3-Month Follow-Up
Changes in Ability to Distancing From Emotional Experience: Experiences Questionnaire (EQ) | Pre-Training, Post-Training (6 weeks after starting the training), and 3-Month Follow-Up
Changes in Ability to Regulate Attention: Attentional Control Scale (ACS) | Pre-Training, Post-Training (6 weeks after starting the training), and 3-Month Follow-Up
Changes in Ability to Regulate Attention in Emotional Contexts: Emotional Attentional Control Scale (eACS) | Pre-Training, Post-Training (6 weeks after starting the training), and 3-Month Follow-Up
Changes in Approach-Avoidance Motivation: Mental Representation of Approach Avoidance Questionnaire (MRAAQ) | Pre-Training, Post-Training (6 weeks after starting the training), and 3-Month Follow-Up
Changes in Positive and Negative Emotions: Modified Differential Emotions Scale (mDES) | Pre-Training, Post-Training (6 weeks after starting the training), and 3-Month Follow-Up
Change in Behavioral Dysregulation: Behavioral Dysregulation Scale (BDRS) | Pre-Training, Post-Training (6 weeks after starting the training), and 3-Month Follow-Up

SECONDARY OUTCOMES:
Changes in Mood and Anxiety Symptoms: Mood and Anxiety Symptoms Questionnaire (MASQ-90) | Pre-Training, Post-Training (6 weeks after starting the training), and 3-Month Follow-Up
Changes in Rumination: Rumination-Reflection Questionnaire (RRQ) | Pre-Training, Post-Training (6 weeks after starting the training), and 3-Month Follow-Up
Changes in Worry: Penn State Worry Questionnaire (PSWQ) | Pre-Training, Post-Training (6 weeks after starting the training), and 3-Month Follow-Up
Changes in Self-Criticism: Self-Judgement Subscale of the Self-Compassion Scale (SCS) | Pre-Training, Post-Training (6 weeks after starting the training), and 3-Month Follow-Up
Changes in Functional Impairment: Sheehan Disability Scale (SDS) | Pre-Training, Post-Training (6 weeks after starting the training), and 3-Month Follow-Up
Changes in Life Satisfaction: Brief Multidimensional Students' Life Satisfaction Scale (BMSLSS) | Pre-Training, Post-Training (6 weeks after starting the training), and 3-Month Follow-Up
Changes in Valued Living/Action: Valuing Questionnaire (VQ) | Pre-Training, Post-Training (6 weeks after starting the training), and 3-Month Follow-Up
Satisfaction and Usability of Treatment: Client Satisfaction Questionnaire (CSQ) | Post-Training (6 weeks after starting the training)

CONTACTS AND LOCATIONS:
Overall Officials: Douglas S Mennin, PhD, Principal Investigator — Teachers College, Columbia University
Locations (1):
- Teachers College, Columbia University, New York, New York, United States